CLINICAL TRIAL: NCT00186888
Title: Protocol for the Study and Treatment of Patients With Intraocular Retinoblastoma
Brief Title: Study of Treatment for Patients With Cancer of the Eye -Retinoblastoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RET5; P01CA023099 (NIH); NCI-2011-01186 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2011-08-30 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Retinoblastoma; Retinal Neoplasm
Keywords: Cancer of the Eye; Eye Enucleation
MeSH Terms: conditions — Retinoblastoma; Retinal Neoplasms; Eye Neoplasms | interventions — Eye Enucleation; Vincristine; Carboplatin; Topotecan; Etoposide; Cyclophosphamide; Doxorubicin; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Stratum A (Other): Patients with early bilateral or unilateral, or patients with bilateral that have already had the advanced eye enucleated. Treatment included vincristine and carboplatin for 8 courses, given at 3-4 week intervals. Focal therapies any time after second course can include cryotherapy, laser photocoagulation, thermotherapy, and plaque radiotherapy
  Interventions: Procedure: Enucleation; Drug: Vincristine, Carboplatin; Procedure: Focal Therapies; Radiation: External Beam Radiation; Other: G-CSF
- Stratum B (Other): Patients with bilateral disease (at least one advanced stage eye), candidate for conservative management.
  Treatment included window treatment with vincristine and topotecan, Followed by 3 more courses of vincristine-topotecan if they had a response to the window+ 6 courses of vincristine and carboplatin. If they do not respond to the window, they receive 6 courses of vincristine, carboplatin, and etoposide. Periocular carboplatin is also given three times, depending on whether they respond to window. External Beam Radiation 44-46 Gy administered using standard practices.
  Interventions: Procedure: Enucleation; Drug: Vincristine, Carboplatin; Procedure: Focal Therapies; Radiation: External Beam Radiation; Drug: Vincristine and Topotecan; Drug: Vincristine + Carboplatin + Etoposide; Procedure: Periocular carboplatin; Other: G-CSF
- Stratum C (Other): Patients with advanced unilateral advanced intraocular disease. First intervention is enucleation.
  If enucleated eye does not have disease outside the retina (low risk), no additional treatment is given.
  For patients whose enucleated eye shows tumor outside the retina (intermediate risk), they will receive 4 courses of vincristine, cyclophosphamide, and doxorubicin followed by G-CSF.
  For patients with high risk disease (involvement of the sclera, optic nerve at the level of the cut-end), treatment after enucleation is 6 courses of alternating chemotherapy with vincristine, carboplatin, etoposide (VCE) to alternate with vincristine, cyclophosphamide, and doxorubicin (VCD). High risk patients also receive external-beam radiation therapy.
  Interventions: Procedure: Enucleation; Radiation: External Beam Radiation; Drug: vincristine, cyclophosphamide, and doxorubicin; Drug: Vincristine, Carboplatin and Etoposide; Other: G-CSF

INTERVENTIONS:
Procedure: Enucleation — Enucleation (possibly associated with all treatment strata/arms. For Stratum A, patients with bilateral disease will have surgery to remove the advanced eye before chemotherapy, or patients that have disease progression after chemotherapy may have surgery to remove the affected eye.
  For Stratum B, Surgical removal of the affected eye may be required in cases of disease progression For Stratum C, first intervention is removal of the affected eye.
Drug: Vincristine, Carboplatin — (Stratum A subjects receive 8 courses every 3-4 weeks, Stratum B subjects receive this combination for Courses 3, 4, 6, 7, 9, and 10 after the window, if they respond to window therapy) Vincristine dosage< 12 months of age: 0.05 mg/kg i.v. day 1, ≥ 12 months of age: 1.5 mg/m2 i.v. day 1 (max. dose 2 mg) Carboplatin will be administered i.v. to achieve an AUC of 6.5 mg/ml/min, day 1.
  Other Names: Oncovin + Paraplatin
  Arms: Stratum A; Stratum B
Procedure: Focal Therapies — Method will be at the discretion of the treating team, used after second course of chemotherapy. Cryotherapy- freezing of affected tissue, Laser photocoagulation- using lasers to destroy affected tissue, Thermotherapy and thermochemotherapy- using heat or heat/chemotherapy combination to destroy diseased tissue, and Episcleral plaque brachytherapy- radiation insertions in the diseased area to destroy affected tissue.
  Arms: Stratum A; Stratum B
Radiation: External Beam Radiation — 44-46 Gy administered using standard practices , limiting dose to normal tissues to subjects with recurrent or progressive disease not considered controllable with focal treatments, Stratum B subjects with suspected active disease after completing therapy, or patients considered to have high-risk disease.
Drug: Vincristine and Topotecan — (Stratum B subjects receive two up-front courses of vincristine and topotecan, given in 21-day intervals, then those who respond receive 3 additional courses (courses 5, 8, and 11) after the window. Dosages are the same for both window and subsequent courses: Vincristine: < 12 months of age: 0.05 mg/kg i.v. day 1, ≥ 12 months of age: 1.5 mg/m2 i.v. day 1 (max. dose 2 mg) Topotecan: TSE of 140 ± 20 ng/ml*hr, daily for 5 consecutive days, infused over 30 minutes.
  Other Names: Oncovin + Hycamtin
  Arms: Stratum B
Drug: Vincristine + Carboplatin + Etoposide — Stratum B patients that do not respond to window receive 6 courses of this combination.
  Vincristine: < 12 months of age: 0.05 mg/kg i.v. day 1, ≥ 12 months of age: 1.5 mg/m2 i.v. day 1 (max. dose 2 mg) Carboplatin will be administered i.v. to achieve an AUC of 6.5 mg/ml/min, day 1 Etoposide, < 12 months of age: 3.3 mg/kg/d i.v. days 1 - 3, ≥ 12 months of age: 100 mg/m2/d i.v. days 1 - 3
  Other Names: Oncovin + Paraplatin + VP-16
  Arms: Stratum B
Drug: vincristine, cyclophosphamide, and doxorubicin — (High risk Stratum C patients in courses 2, 4, and 6 after enucleation, intermediate risk stratum C patients for four consecutive courses after enucleation) Vincristine: < 12 months of age: 0.05 mg/kg i.v. day 1, ≥ 12 months of age: 1.5 mg/m2 i.v. day 1 (max. dose 2 mg) Cyclophosphamide: < 12 months of age: 40 mg/kg i.v. day 1, ≥ 12 months of age: 1,200 mg/m2 i.v. day 1, MESNA 200 mg/m2 at 0, 3, 6, and 9 hours Doxorubicin < 12 months of age: 1.5 mg/kg i.v. day 1, ≥ 12 months of age: 45 mg/m2 i.v. day 1
  Other Names: Onconvin and Cytoxan and Adriamycin
  Arms: Stratum C
Drug: Vincristine, Carboplatin and Etoposide — High risk Stratum C patients in courses 1, 3, and 5 after enucleation: Vincristine: < 12 months of age: 0.05 mg/kg i.v. day 1, ≥ 12 months of age: 1.5 mg/m2 i.v. day 1 (max. dose 2 mg) Carboplatin will be administered i.v. to achieve an AUC of 6.5 mg/ml/min, day 1 Etoposide, < 12 months of age: 3.3 mg/kg/d i.v. days 1 - 3, ≥ 12 months of age: 100 mg/m2/d i.v. days 1 - 3
  Other Names: Onconvin and Paraplatin and Vepesid
  Arms: Stratum C
Procedure: Periocular carboplatin — Periocular (subtenon) carboplatin 20 mg, one injection, in courses 5, 8, and 11 in patients responding to the VT window, and in courses 1, 3, and 6 of VCE in patients not responding to the VT window, when active vitreous disease is present. Carboplatin 20 mg will be diluted in 2 mL of NS or D5W and given by subtenon administration while the patient is under general anesthesia.
  Other Names: Paraplatin
  Arms: Stratum B
Other: G-CSF — G-CSF (5 mcg/kg/day), will be administered starting 24-36 hours after the completion of each course of chemotherapy, for 7 to 10 days, until ANC is > 2,000/mL in one occasion after the expected nadir.
  Other Names: Filgrastim; Neupogen

SUMMARY:
Retinoblastoma is a childhood cancer which affects the retina of the eye. The retina is the light sensitive layer of tissue that lines the back of the eyeball; sends visual messages through the optic nerve to the brain. When only one eye is affected, this is known as unilateral retinoblastoma and when both eyes are affected, it is called bilateral retinoblastoma. Treatment for retinoblastoma is individualized for each patient and is based on the form and the stage of the disease (inside the eye or has moved outside). The main goal is always to cure the cancer, and save the life of the child. Treatments are also designed with the hope of saving the vision, while completely destroying the tumor. Therapies may involve surgery, chemotherapy, radiation, and other treatments called focal treatments. Focal treatments may be laser therapy, freezing, or heat treatments meant to shrink and kill the tumor.

In this study, researchers want to investigate how different participants respond to different therapies that are individualized specifically for them. Participants will be divided into three main groups, depending on whether the disease is unilateral or bilateral, and the stage of the disease. One of the main objectives of the study is to investigate how advanced tumors in children with bilateral disease respond to a new combination of chemotherapy with topotecan and vincristine, with G-CSF support. In order to improve results, some children with very advanced disease may receive carboplatin chemotherapy given around the eye at the same time that they receive topotecan by vein. Also, because children with retinoblastoma are diagnosed so early in life and the vision may be significantly impaired, this study will investigate how children develop and how the brain adjusts and compensates for the visual deficits. Finally, this study also investigates the biology of retinoblastoma, in order to understand better how this cancer develops.

DETAILED DESCRIPTION:
This study will determine the following:

PRIMARY OBJECTIVE:

* To estimate the ocular survival and event-free survival of bilateral disease patients with advanced intraocular retinoblastoma in either eye (R-E IV-V) responding to the vincristine/topotecan window, with alternating cycles of vincristine and carboplatin with vincristine, topotecan, and periocular carboplatin, with intensive focal treatments.

SECONDARY OBJECTIVES:

* To estimate the ocular survival of eye and event-free survival of eye of bilateral disease patients with advanced intraocular retinoblastoma in either eye (R-E IV-V) responding to the vincristine/topotecan window, with alternating cycles of vincristine and carboplatin with vincristine, topotecan, and periocular carboplatin, with intensive focal treatments.
* To estimate the ocular survival and event free survival of patients with advanced intraocular retinoblastoma (R-E IV-V) not responding to the vincristine/topotecan window, with a combination of vincristine, carboplatin, etoposide, and periocular carboplatin, with intensive focal treatments.
* To estimate the ocular survival and event free survival of eye of patients with advanced intraocular retinoblastoma (R-E IV-V) not responding to the vincristine/topotecan window, with a combination of vincristine, carboplatin, etoposide, and periocular carboplatin, with intensive focal treatments.
* To estimate the ocular survival and event-free survival of patients with early stage intraocular retinoblastoma (R-E I-III) with vincristine and carboplatin with intensive focal treatments.
* To estimate the ocular survival of eye and event-free survival of eye of patients with early stage intraocular retinoblastoma (R-E I-III) with vincristine and carboplatin with intensive focal treatments.
* To estimate the response rate of early stage eyes (R-E I-III) in patients with contralateral advanced disease treated with vincristine and topotecan.
* To estimate the ocular survival and event-free survival of early stage eyes (R-E I-III) of patients with contralateral advanced disease treated with vincristine and topotecan.
* To describe the outcome of intraocular retinoblastoma with respect to the new International Classification for Intraocular Retinoblastoma and the AJCC.
* To describe primary visual cortex function in patients with unilateral and bilateral retinoblastoma.
* To describe the cognitive, adaptive, and social/emotional development of children with retinoblastoma.
* To describe changes in the pineal gland during treatment in patients with bilateral retinoblastoma.
* To assess the relation between CYP3A4/5 genotype and the pharmacokinetics and pharmacodynamics of topotecan.
* To assess the relation between ABCG2 genotype and the pharmacokinetics and pharmacodynamics of topotecan.
* To determine if carboplatin can produce changes in cochlear function that are detectable with measurement of otoacoustic emissions.
* To evaluate the need for and feasibility of starting early intervention support during the first year after the diagnosis of retinoblastoma.

EXPLORATORY OBJECTIVES:

* To provide insight into molecular pathogenesis of retinoblastoma.
* To describe the incidence and type of germline mutations of the RB gene in patients with retinoblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Must have newly diagnosed intraocular retinoblastoma, previously untreated. Patients previously diagnosed with unilateral retinoblastoma treated surgically (or with focal therapies), who develop asynchronous involvement of the contralateral eye, will be eligible for study.
* Must have a life expectancy of at least 8 weeks.
* Must have Performance Status (ECOG) of 0-2.
* Patients must have an adequate liver function, as defined by bilirubin less than or equal to 3 x normal, and SGOT and SGPT less than or equal to 3x normal.
* Patients must have adequate renal function as defined by serum creatinine less than or equal to 3x normal for age.
* Legal guardians must sign an informed consent indicating that they are aware of this study, its possible benefits, and toxic side effects. Legal guardians will be given a copy of the consent form.

Exclusion Criteria:

* Previously treated patients
* Presence of metastatic disease or orbital involvement
* Patients must not have an invasive infection at time of protocol entry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2005-04-07 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2024-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Qaddoumi, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] King BA, Sahr N, Sykes A, Wilson MW, Brennan RC. Chemoreduction with topotecan and vincristine: Quantifying tumor response in bilateral retinoblastoma patients. Pediatr Blood Cancer. 2021 Apr;68(4):e28882. doi: 10.1002/pbc.28882. Epub 2021 Jan 28. PMID 33507604
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 107 patients were recruited between February, 2005 and June, 2010 (stratum B) and between February, 2005 and November, 2010 (strata A & C).The primary objective was designed only for stratum B patients who had advanced bilateral retinoblastoma and received the investigational window therapy.
Pre-assignment Details: 107 patients were enrolled on the study. Two patients were excluded as they were deemed to be ineligible after study enrollment. One patient was found to have retinal dysplasia rather than retinoblastoma and the other patient had retinoblastoma but did not fit into any of the defined treatment strata for this study.
Groups:
- Stratum A: Early Unilateral or Bilateral Retinoblastoma. Stratum A includes mainly patients with early stage (Reese-Ellsworth group I, II, or III) bilateral retinoblastoma. Patients with unilateral disease diagnosed at an early stage, and patients with early multifocal unilateral disease are rare, but these patients are also candidates for conservative management and were treated in stratum A.
- Stratum B: Advanced Bilateral Retinoblastoma. Stratum B includes patients with at least one Reese-Ellsworth group IV or V eye that after careful evaluation by the treating team is considered not to require upfront enucleation. A proportion of patients treated on this stratum will not have advanced disease in both eyes. Only stratum B patients received window therapy consisting of 2 courses of vincristine and topotecan.
- Stratum C: Advanced Unilateral Retinoblastoma. Research participants with unilateral (unifocal or multifocal) advanced (Reese-Ellsworth group IV or V) intraocular disease will undergo upfront enucleation. Adjuvant therapy was also indicated in certain cases.
Period: Overall Study
Arm/Group | Stratum A | Stratum B | Stratum C
Started | 23 | 27 | 55
Window Therapy | 0 | 27 | 0
Completed | 19 | 24 | 55
Not Completed | 4 | 3 | 0
Not completed — Toxicity | 0 | 1 | 0
Not completed — Relapse or progression of disease | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum A | Stratum B | Stratum C | Total
Number analyzed (Participants) | 23 | 27 | 55 | 105
Age, Continuous [Mean (Standard Deviation); unit: months] | 5.7 (3.6) | 8.5 (4.6) | 29.6 (22.1) | 18.9 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 28 | 52
  Male | 12 | 14 | 27 | 53
Tumor Laterality [Count of Participants; unit: Participants] — Population: Evaluable visual cortex (V1) activation for longitudinal analysis was detected in 77 patients.
  Participants
    number analyzed (Participants) | 12 | 24 | 41 | 77
    Bilateral Tumor | 3 | 24 | 0 | 27
    Unilateral Tumor | 9 | 0 | 41 | 50

OUTCOME MEASURES:

1. Primary Outcome: Stratum B Response to Window Therapy
Description: The primary outcome is to estimate the proportion of stratum B patients responding to 2 courses of window therapy consisting of vincristine and topotecan. Complete Response is the complete regression of all apparent tumor masses in the funduscopic examination and by MRI and ultrasound (US). Partial Response is defined as greater than 50% (but less than 100%) reduction of the tumor masses in the funduscopic examination and by US and MRI, without the appearance of any new lesions. The response must persist for at least 4 weeks. Stratum A and C did not receive window therapy.
Time Frame: Six weeks post window therapy
Population: The primary objective related to stratum B patients only, as these were the patients who were given window therapy consisting of 2 courses of vincristine and topotecan. Of the 27 stratum B patients enrolled, all were included in the analysis of the primary objective.
Measure: Number; unit: Participants
Arm/Group | Stratum B
Number analyzed (Participants) | 27
Participants
  Partial response | 24
  Progressive Disease or New Lesion | 2
  Failure due to Toxicity | 1
Statistical Analysis 1: Comparison: Stratum B; Test type: Superiority or Other; Binomial Proportion = 88.9, 95% CI 2-sided [71.3 to 96.9]

2. Secondary Outcome: Stratum B Response Rate of Early Stage Eyes to Window Therapy
Description: To estimate the proportion of early stage eyes defined as Reese-Ellsworth Group I, II, or III eyes, that responded to 2 courses of window therapy which consisted of vincristine and topotecan
Time Frame: Six weeks post window therapy.
Population: Among the 27 stratum B patients with 54 eyes with retinoblastoma, 12 eyes were early stage (Reese-Ellsworth group I, II, or III). The remaining 42 eyes were advanced stage and were not included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Stratum B
Number analyzed (Participants) | 12
Participants
  Partial response | 11
  Progressive Disease / New lesion | 0
  Failure due to Toxicity | 1
Statistical Analysis 1: Comparison: Stratum B; Test type: Superiority or Other; Binomial Proportion = 91.7, 95% CI 2-sided [65.1 to 99.6]

3. Secondary Outcome: Relationship Between Topotecan Clearance (CL) and CYP3A4/5 Genotype in Stratum B Participants.
Description: Blood samples for pharmacokinetic studies were collected at 0 hour (pre-dose), 5 minutes, 1.5 and 2.5 hours after the end of topotecan dose on Course 1 Day 1, Course 2 Day 1, and if further studies were needed, Course 5 Day 1 and Course 8 Day 1. A blood sample for pharmacogenetic studies was collected during the course of therapy on protocol.
Time Frame: Courses 1, 2, 5, and 8
Population: Of the 107 participants enrolled in the overall study, analysis was performed for 19 participants who were enrolled on Stratum B AND who had results for both topotecan clearance and pharmacogenetic studies.
  Only wild-type was present in CYP3A5*6, therefore, statistical analysis was not done for these alleles.
Measure: Median (95% Confidence Interval); unit: Liters/hour/m^2
Arm/Group | Stratum B
Number analyzed (Participants) | 19
Liters/hour/m^2 | 18.8 [9.8 to 36.8]
Statistical Analysis 1: Comparison: Stratum B; CYP3A4*1B: The null hypothesis is there is not a statistically significant difference between the genotype groups; Test type: Superiority or Other; p = 0.452, ANOVA
Statistical Analysis 2: Comparison: Stratum B; CYP3A5*3: The null hypothesis is there is not a statistically significant difference between the genotype groups; Test type: Superiority or Other; p = 0.106, ANOVA

4. Secondary Outcome: Relationship Between Topotecan Clearance (CL) and ABCG2/B1 Genotype in Stratum B Participants.
Description: as for outcome 3
Time Frame: Courses 1, 2, 5, and 8
Population: Of the 107 participants enrolled in the overall study, analysis was performed for 19 participants who were enrolled on Stratum B AND who had results for both topotecan clearance and pharmacogenetic studies.
  Only wild-type was present in BCRP 15994, therefore, statistical analysis was not done for these alleles.
Measure: Median (95% Confidence Interval); unit: Liters/hour/m^2
Arm/Group | Stratum B
Number analyzed (Participants) | 19
Liters/hour/m^2 | 18.8 [9.8 to 36.8]
Statistical Analysis 1: Comparison: Stratum B; BCRP 1143: The null hypothesis is there is not a statistically significant difference between the genotype groups; Test type: Superiority or Other; p = 0.245, ANOVA
Statistical Analysis 2: Comparison: Stratum B; BCRP 15622: The null hypothesis is there is not a statistically significant difference between the genotype groups; Test type: Superiority or Other; p = 0.297, ANOVA
Statistical Analysis 3: Comparison: Stratum B; BCRP Exon 2: The null hypothesis is there is not a statistically significant difference between the genotype groups; Test type: Superiority or Other; p = 0.372, ANOVA
Statistical Analysis 4: Comparison: Stratum B; BCRP Exon 5: The null hypothesis is there is not a statistically significant difference between the genotype groups; Test type: Superiority or Other; p = 0.844, ANOVA
Statistical Analysis 5: Comparison: Stratum B; Pgp Exon 21: The null hypothesis is there is not a statistically significant difference between the genotype groups; Test type: Superiority or Other; p = 0.616, ANOVA
Statistical Analysis 6: Comparison: Stratum B; Pgp Exon 26: The null hypothesis is there is not a statistically significant difference between the genotype groups; Test type: Superiority or Other; p = 0.424, ANOVA

5. Secondary Outcome: Event-free Survival of Stratum B Patients Responding to Window Treatment
Description: To estimate the 5-year event-free (EFS) survival of bilateral disease patients with advanced intraocular retinoblastoma in either eye (R-E IV-V) responding to the vincristine/topotecan window, with alternating cycles of vincristine and carboplatin with vincristine, topotecan, and periocular carboplatin, with intensive focal treatments.
  Event-free survival will be defined per patient as follows: for patients with one advanced stage eye, the time interval from date on study to date of first event (an event includes external beam radiation or enucleation) of advanced stage eyes, time to first event will be used for the analysis. Event-free survival will be estimated using the method of Kaplan and Meier.
Time Frame: From date on-study to an event or last follow-up
Population: Of the total 27 eligible patients in stratum B, 3 patients were not responding to the window therapy; 1 withdrew the consent and was taken off the study, and 2 developed disease progression. Kaplan and Meier estimate of ocular survival was calculated for the remaining 24 patients.
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- Stratum B: Advanced Bilateral Retinoblastoma. Stratum B includes patients with at least one Reese-Ellsworth group IV or V eye that after careful evaluation by the treating team is considered not to require upfront enucleation. A proportion of patients treated on this stratum will not have advanced disease in both eyes. Only stratum B patients received window therapy consisting of 2 courses of vincristine and topotecan.
  Two patients (3 eyes) in stratum B received external beam radiation therapy (EBRT), and the same 2 patients later required enucleation of the treated eye, thus the failure (event number) and censoring status were not changed for the 2 patients.
Arm/Group | Stratum B
Number analyzed (Participants) | 24
probability | 0.667 [0.478 to 0.855]

6. Secondary Outcome: Ocular Survival of Stratum B Patients Responding to Window Treatment
Description: To estimate the 5-year ocular survival of bilateral disease patients with advanced intraocular retinoblastoma in either eye (R-E IV-V) responding to the vincristine/topotecan window, with alternating cycles of vincristine and carboplatin with vincristine, topotecan, and periocular carboplatin, with intensive focal treatments.
  Ocular survival will be defined per patient as follows: for patients with one advanced stage eye, the time interval from date on study to date of enucleation of advanced stage eye or date of last follow-up, for patients with two advanced stage eyes, the time to the first enucleation will be used for analysis. Ocular survival will be estimated using the method of Kaplan and Meier. Standard error is 5-year ocular survival
Time Frame: From date on-study to an event or last follow-up
Population: From the total of 27 eligible patients in stratum B, 3 patients were not responding to the window therapy; 1 withdrew the consent and was taken off the study, and 2 developed disease progression. Thus, the Kaplan and Meier estimate of ocular survival was calculated for the remaining 24 patients.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Stratum B
Number analyzed (Participants) | 24
probability | 0.667 [0.478 to 0.855]

7. Secondary Outcome: Event-free Survival of Eyes in Stratum B Patients Responding to Window Treatment
Description: To estimate the 5-year event-free survival (EFS) of eyes of bilateral disease patients with advanced intraocular retinoblastoma in either eye (R-E IV-V) responding to the vincristine/topotecan window, with alternating cycles of vincristine and carboplatin with vincristine, topotecan, and periocular carboplatin, with intensive focal treatments.
  Event-free survival of eye will be defined per eye as the time interval from date on study to date of first event (an event includes external beam radiation or enucleation) or to last follow-up date for eyes without events. Event-free survival of eye will be estimated using the method of Kaplan and Meier. Standard error is 5-year EFS.
Time Frame: From date on-study to an event or last follow-up
Population: Of the 52 eyes (26 evaluable patients), 2 eyes (2 patients) were removed from analysis as they were not responsive to window therapy. In both cases, the contralateral eye was included in the analysis. One patient with upfront enucleation had only one eye for analysis. Eleven eyes were R-E Group I-III and were excluded. Total: 38 eyes for analysis.
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: Eyes
Arm/Group | Stratum B
Number analyzed (Participants) | 25
Number analyzed (Eyes) | 38
probability | 0.763 [0.628 to 0.898]

8. Secondary Outcome: Ocular Survival of Eyes in Stratum B Patients Responding to Window Treatment
Description: To estimate the 5-year ocular survival of eye of bilateral disease patients with advanced intraocular retinoblastoma in either eye (R-E IV-V) responding to the vincristine/topotecan window, with alternating cycles of vincristine and carboplatin with vincristine, topotecan, and periocular carboplatin, with intensive focal treatments.
  Ocular survival of eye will be defined per eye as the time interval from date on study to date of enucleation or date of last follow-up. Ocular survival of eye will be estimated using the method of Kaplan and Meier. Standard error is 5-year ocular survival.
Time Frame: From date on-study to an event or last follow-up
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: Eyes
Arm/Group | Stratum B
Number analyzed (Participants) | 25
Number analyzed (Eyes) | 38
probability | 0.763 [0.628 to 0.898]

9. Secondary Outcome: Event-free Survival of Stratum B Patients Not Responding to Window Treatment
Description: To estimate the 5-year event free survival of patients with advanced intraocular retinoblastoma (R-E IV-V) not responding to the vincristine/topotecan window, with a combination of vincristine, carboplatin, etoposide, and periocular carboplatin, with intensive focal treatments.
Time Frame: From date on-study to an event or last follow-up
Population: The study closed to enrollment early due to poor accrual, but it remains open to follow-up. Both patients who developed new lesions in one eye during window therapy had a good response in the contralateral eye, and they continued on protocol therapy with vincristine/topotecan. Therefore, no patients were treated with this combination therapy.
Arm/Group | Stratum B
Number analyzed (Participants) | 0

10. Secondary Outcome: Ocular Survival of Stratum B Patients Not Responding to Window Treatment
Description: To estimate the 5-year ocular survival of patients with advanced intraocular retinoblastoma (R-E IV-V) not responding to the vincristine/topotecan window, with a combination of vincristine, carboplatin, etoposide, and periocular carboplatin, with intensive focal treatments.
Time Frame: From date on-study to an event or last follow-up
Population: as for outcome 9
Arm/Group | Stratum B
Number analyzed (Participants) | 0

11. Secondary Outcome: Event-free Survival of Eyes in Stratum B Patients Not Responding to Window Treatment
Description: To estimate the 5-year event free survival of the eye of patients with advanced intraocular retinoblastoma (R-E IV-V) not responding to the vincristine/topotecan window, with a combination of vincristine, carboplatin, etoposide, and periocular carboplatin, with intensive focal treatments
Time Frame: From date on-study to an event or last follow-up
Population: as for outcome 9
Arm/Group | Stratum B
Number analyzed (Participants) | 0

12. Secondary Outcome: Ocular Survival of Eyes in Stratum B Patients Not Responding to Window Treatment
Description: To estimate the 5-year ocular survival of the eye of patients with advanced intraocular retinoblastoma (R-E IV-V) not responding to the vincristine/topotecan window, with a combination of vincristine, carboplatin, etoposide, and periocular carboplatin, with intensive focal treatments
Time Frame: From date on-study to an event or last follow-up
Population: as for outcome 9
Arm/Group | Stratum B
Number analyzed (Participants) | 0

13. Secondary Outcome: Event-free Survival of Stratum A Patients
Description: To estimate the 5-year event-free survival of patients with early stage intraocular retinoblastoma (R-E I-III) with vincristine and carboplatin with intensive focal treatments.
  Event-free survival will be defined per patient as follows: for patients with one advanced stage eye, the time interval from date on study to date of first event (an event includes external beam radiation or enucleation) of advanced stage eyes, time to first event will be used for the analysis. Event-free survival will be estimated using the method of Kaplan and Meier.
Time Frame: From date on-study to an event or last follow-up
Population: All 23 stratum A patients received VC treatment and focal therapy.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Stratum A
Number analyzed (Participants) | 23
probability | 0.688 [0.496 to 0.880]

14. Secondary Outcome: Ocular Survival of Stratum A Patients
Description: To estimate the 5-year ocular survival of patients with early stage intraocular retinoblastoma (R-E I-III) with vincristine and carboplatin with intensive focal treatments.
  Ocular survival will be defined per patient as follows: for patients with one advanced stage eye, the time interval from date on study to date of enucleation of advanced stage eye or date of last follow-up, for patients with two advanced stage eyes, the time to the first enucleation will be used for analysis. Ocular survival will be estimated using the method of Kaplan and Meier.
Time Frame: From date on-study to an event or last follow-up
Population: All 23 stratum A patients received VC treatment and focal therapy.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Stratum A
Number analyzed (Participants) | 23
probability | 0.688 [0.496 to 0.880]

15. Secondary Outcome: Event-free Survival of Eyes of Stratum B Patients
Description: To estimate the 5-year event-free survival of early stage eyes (R-E I-III) of patients with contralateral advanced disease treated with vincristine and topotecan.
  Event-free survival of eye will be defined per eye as the time interval from date on study to date of first event (an event includes external beam radiation or enucleation) or to last follow-up date for eyes without events. Event-free survival of eye will be estimated using the method of Kaplan and Meier.
Time Frame: From date on-study to an event or last follow-up
Population: The criteria considered eyes of all stratum B patients with R-E I-III (11 eyes in 11 patients).
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: Eyes
Arm/Group | Stratum B
Number analyzed (Participants) | 11
Number analyzed (Eyes) | 11
probability | 1.0 [NA to NA] — There is no event in the data, thus SE=0 and 95% CI is not available.

16. Secondary Outcome: Ocular Survival of Eyes of Stratum B Patients
Description: To estimate the 5-year ocular survival of early stage eyes (R-E I-III) of patients with contralateral advanced disease treated with vincristine and topotecan.
  Ocular survival will be defined per patient as follows: for patients with one advanced stage eye, the time interval from date on study to date of enucleation of advanced stage eye or date of last follow-up, for patients with two advanced stage eyes, the time to the first enucleation will be used for analysis. Ocular survival will be estimated using the method of Kaplan and Meier.
Time Frame: From date on-study to an event or last follow-up
Population: The criteria considered eyes of all stratum B patients with R-E I-III (11 eyes in 11 patients).
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: Eyes
Arm/Group | Stratum B
Number analyzed (Participants) | 11
Number analyzed (Eyes) | 11
probability | 1.0 [NA to NA] — There is no event in the data, thus SE=0 and 95% CI is not available.

17. Secondary Outcome: Event-free Survival of Eyes in Stratum A and Stratum B Patients Based on IC Classification
Description: To describe the 5-year event-free survival of the eyes outcome of intraocular retinoblastoma with respect to the new International Classification (IC) for Intraocular Retinoblastoma and the AJCC.
  Patients were re-classified into 2 groups of early (IC groups A and B) and advanced (IC groups C, D, and E) retinoblastoma. Analysis was done at eye level since each eye in the same patient could be a different group. Patients from stratum A and B were analyzed separately.
  Three eyes (2 patients) in stratum B received external beam radiation therapy (EBRT) and were also coincident with enucleation surgery, so their event status was not changed. Although the 3 eyes had shorter EFS interval because EBRT occurred (less than 2 years) before the surgery, it did not change the 5-year survival probability.
Time Frame: From date on-study to an event or last follow-up
Population: For the 23 stratum A patients, 35 eyes (12 bilateral patients, 11 unilateral patients) with IC grouping were analyzed. For 26 Stratum B patients, 1 eye with up-front surgery was excluded from analysis. 51 eyes with IC grouping were analyzed. Participants with bilateral disease may have one eye in each category.
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: Number of Eyes
Groups:
- Stratum A-Early Disease; Stratum A-Advanced Disease: Early Unilateral or Bilateral Retinoblastoma. Stratum A includes mainly patients with early stage (Reese-Ellsworth group I, II, or III) bilateral retinoblastoma. Patients with unilateral disease diagnosed at an early stage, and patients with early multifocal unilateral disease are rare, but these patients are also candidates for conservative management and were treated in stratum A.
  The patients were re-classified into 2 groups of early (IC Group=A and B) and advanced (IC Group=C, D, E) retinoblastoma. The analysis was done at eye level since each eye in the same patient could be a different group.
- Stratum B-Early Disease; Stratum B-Advanced Disease: Advanced Bilateral Retinoblastoma. Stratum B includes patients with at least one Reese-Ellsworth group IV or V eye that after careful evaluation by the treating team is considered not to require upfront enucleation. A proportion of patients treated on this stratum will not have advanced disease in both eyes. Only stratum B patients received window therapy consisting of 2 courses of vincristine and topotecan.
  The patients were re-classified into 2 groups of early (IC Group=A and B) and advanced (IC Group=C, D, E) retinoblastoma. The analysis was done at eye level since each eye in the same patient could be a different group.
Arm/Group | Stratum A-Early Disease | Stratum A-Advanced Disease | Stratum B-Early Disease | Stratum B-Advanced Disease
Number analyzed (Participants) | 18 | 9 | 15 | 25
Number analyzed (Number of Eyes) | 26 | 9 | 16 | 35
probability | 0.839 [0.694 to 0.984] | 0.667 [0.359 to 0.975] | 1.0 [NA to NA] — There is no event in the data, thus SE=0 and 95% CI is not available. | 0.743 [0.598 to 0.888]

18. Secondary Outcome: Ocular Survival of Eyes in Stratum A and Stratum B Patients Based on IC Classification
Description: To describe the 5-year ocular survival of eyes outcome of intraocular retinoblastoma with respect to the new International Classification (IC) for Intraocular Retinoblastoma and the AJCC.
  Patients were re-classified into 2 groups of early (IC groups A and B) and advanced (IC groups C, D, and E) retinoblastoma. Analysis was done at eye level since each eye in the same patient could be a different group. Patients from stratum A and B were analyzed separately.
  Three eyes (2 patients) in stratum B received external beam radiation therapy (EBRT) and were also coincident with enucleation surgery, so their event status was not changed. Although the 3 eyes had shorter EFS interval because EBRT occurred (less than 2 years) before the surgery, it did not change the 5-year survival probability.
Time Frame: From date on-study to an event or last follow-up
Population: For the 23 stratum A patients, 35 eyes (12 bilateral patients, 11 unilateral patients) with IC grouping were analyzed.For 26 Stratum B patients, 1 eye with up-front surgery was excluded from analysis. 51 eyes with IC grouping were analyzed. Participants with bilateral disease may have one eye in each category.
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: Eyes
Groups:
- Stratum A-Advanced Disease: Early Unilateral or Bilateral Retinoblastoma. Stratum A includes mainly patients with early stage (Reese-Ellsworth group I, II, or III) bilateral retinoblastoma. Patients with unilateral disease diagnosed at an early stage, and patients with early multifocal unilateral disease are rare, but these patients are also candidates for conservative management and were treated in stratum A.
  The patients were re-classified into 2 groups of early (IC=A and B) and advanced (IC=C, D, E) retinoblastoma. The analysis was done at eye level since each eye in the same patient could be a different group.
Arm/Group | Stratum A-Early Disease | Stratum A-Advanced Disease | Stratum B-Early Disease | Stratum B-Advanced Disease
Number analyzed (Participants) | 18 | 9 | 15 | 25
Number analyzed (Eyes) | 26 | 9 | 16 | 35
probability | 0.839 [0.694 to 0.984] | 0.667 [0.359 to 0.975] | 1.0 [NA to NA] — There is no event in the data, thus SE=0 and 95% CI is not available. | 0.743 [0.598 to 0.888]

19. Secondary Outcome: Event-free Survival Per Eye in Stratum A and Stratum B Patients Based on AJCC Classification
Description: To describe the 5-year event-free survival of eyes outcome of intraocular retinoblastoma with respect to the new classification of the American Joint Committee on Cancer (AJCC).
  For AJCC staging, the patients were re-classified into 2 groups of early (AJCC=1, 1a or 1b) and advanced (AJCC=2, 2a, 2b, 3, 3a, 3b) retinoblastoma. The analysis was done at eye level since each eye in the same patient could be a different group. Patients from stratum A and B were analyzed separately
Time Frame: From date on-study to an event or last follow-up
Population: For the 23 stratum A patients, 35 eyes (12 bilateral patients, 11 unilateral patients) with IC grouping were analyzed. For 26 Stratum B patients, 1 eye with up-front surgery was excluded from analysis. Participants with bilateral disease may have one eye in each category.
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: Eyes
Groups:
- Stratum A-Early Disease; Stratum A-Advanced Disease: Early Unilateral or Bilateral Retinoblastoma. Stratum A includes mainly patients with early stage (Reese-Ellsworth group I, II, or III) bilateral retinoblastoma. Patients with unilateral disease diagnosed at an early stage, and patients with early multifocal unilateral disease are rare, but these patients are also candidates for conservative management and were treated in stratum A.
  The patients were re-classified into 2 groups of early (AJCC=1, 1a or 1b) and advanced (AJCC=2, 2a, 2b, 3, 3a, 3b) retinoblastoma. The analysis was done at eye level since each eye in the same patient could be a different group.
- Stratum B-Early Disease; Stratum B-Advanced Disease: Advanced Bilateral Retinoblastoma. Stratum B includes patients with at least one Reese-Ellsworth group IV or V eye that after careful evaluation by the treating team is considered not to require upfront enucleation. A proportion of patients treated on this stratum will not have advanced disease in both eyes. Only stratum B patients received window therapy consisting of 2 courses of vincristine and topotecan.
  The patients were re-classified into 2 groups of early (AJCC=1, 1a or 1b) and advanced (AJCC=2, 2a, 2b, 3, 3a, 3b) retinoblastoma. The analysis was done at eye level since each eye in the same patient could be a different group.
Arm/Group | Stratum A-Early Disease | Stratum A-Advanced Disease | Stratum B-Early Disease | Stratum B-Advanced Disease
Number analyzed (Participants) | 19 | 6 | 18 | 25
Number analyzed (Eyes) | 29 | 6 | 19 | 32
probability | 0.857 [0.726 to 0.987] | 0.500 [0.100 to 0.900] | 1.0 [NA to NA] — There is no event in the data, thus SE=0 and 95% CI is not available. | 0.719 [0.563 to 0.875]

20. Secondary Outcome: Ocular Survival Per Eye in Stratum A and Stratum B Patients Based on AJCC Classification
Description: To describe the 5-year ocular survival of eyes outcome of intraocular retinoblastoma with respect to the new classification of the American Joint Committee on Cancer (AJCC).
  For AJCC staging, the patients were classified into 2 groups of early (AJCC=1, 1a or 1b) and advanced (AJCC=2, 2a, 2b, 3, 3a, 3b) retinoblastoma . The analysis was done at eye level since each eye in the same patient could be a different group. Patients from stratum A and B were analyzed separately
Time Frame: From date on-study to an event or last follow-up
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: probability
Units Other Than Participants: Number of Eyes
Arm/Group | Stratum A-Early Disease | Stratum A-Advanced Disease | Stratum B-Early Disease | Stratum B-Advanced Disease
Number analyzed (Participants) | 19 | 6 | 18 | 25
Number analyzed (Number of Eyes) | 29 | 6 | 19 | 32
probability | 0.857 [0.726 to 0.987] | 0.500 [0.100 to 0.900] | 1.0 [NA to NA] — There is no event in the data, thus SE=0 and 95% CI is not available. | 0.719 [0.563 to 0.875]

21. Secondary Outcome: Change in Cognitive Functioning
Description: The Early Learning Composite was assessed with Mullen Scales of Early Learning, a measure of developmental functioning appropriate for use with children from birth through age 5. It is an examiner-administered instrument that uses toys, games, pictures, and other objects to elicit information about a child's language, fine and gross motor skills, and overall early learning capabilities. Raw scores are converted to an age-normed standard score (normative mean = 100, SD = 15) for the overall Early Learning Composite. This measure was given at all time points. Higher scores are indicative of better functioning, with scores from 85-115 in the average range.
Time Frame: Baseline (at study entry) and at ages 6 months, 1 year, 2 years, 3 years and 5 years
Population: Data was collected from 94 unique patients. All patients were included, regardless of treatment strata. If the patient age at study entry (baseline) was within the window of an identified time point, their information was included with that time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline: At study entry.
- 6 Months: Participants at 6 months of age ±3 months.
- 1 Year: Participant age was 1 year ±3 months.
- 2 Years: Participant age was 2 years ±3 months.
- 3 Years: Participant age was 3 years ±3 months.
- 5 Years: Participant age was 5 years ±3 months.
Arm/Group | Baseline | 6 Months | 1 Year | 2 Years | 3 Years | 5 Years
Number analyzed (Participants) | 25 | 30 | 50 | 64 | 67 | 60
units on a scale | 91.61 (16.93) | 90.96 (17.66) | 95.91 (17.98) | 88.40 (18.72) | 82.12 (19.75) | 86.00 (15.31)

22. Secondary Outcome: Change in Relevant Daily Living Skills
Description: The Adaptive Behavior composite was measured using the Vineland Scales of Adaptive Behavior (VABS) which is an examiner-administered semi-structured interview that assesses adaptive functioning from birth through adulthood. Subscales including motor skills, communication, socialization, and daily living skills combine into an overall adaptive behavior composite which is an age-normed standard score (normative mean = 100, SD = 15). This measure was given at all time points. Higher scores are indicative of better functioning, with scores from 85-115 in the average range.
Time Frame: Baseline (at study entry), 6 months, 1 year, 2 years, 3 years, and 5 years
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | 6 Months | 1 Year | 2 Years | 3 Years | 5 Years
Number analyzed (Participants) | 25 | 30 | 50 | 64 | 67 | 60
units on a scale | 97.48 (13.35) | 104.73 (11.04) | 106.06 (10.38) | 94.22 (15.44) | 96.45 (19.12) | 93.03 (17.45)

23. Secondary Outcome: Change in Parent Report of Social-Emotional Factors
Description: This outcome was measured using the Ages and Stages Questionnaire which is a parent-completed measure of a child's social-emotional functioning. Raw scores are calculated and compared to cut-off points by age (6 months = 45; 1 year = 48; 2 years = 50; 3 years = 59; 5 years =70). Higher scores are indicative of more problems with scores above the cut-off indicating significant concerns warranting additional follow-up. Possible scores range from 0 to 200+, depending on the number of items administered, which varies by the age of the child (19 to 33 items). However, the primary use of this tool is as a screener. Thus, typically, scores are interpreted as they compare to the identified cut-offs, with children who score above the cut-off referred for further evaluation. This measure was given at all time points.
Time Frame: Baseline (at study entry), 6 months, 1 year, 2 years, 3 years, and 5 years
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | 6 Months | 1 Year | 2 Years | 3 Years | 5 Years
Number analyzed (Participants) | 25 | 30 | 50 | 64 | 67 | 60
units on a scale | 40 (31.12) | 19.42 (14.02) | 26.28 (13.93) | 29.67 (20.83) | 40.61 (37.76) | 39.93 (34.03)

24. Secondary Outcome: Change in Parenting Stress Index (PSI)
Description: The PSI is a commonly used measure of parenting stress. In 101 questions, the PSI delineates between stress as a function of child characteristics (e.g., adaptability, demandingness, mood; Child Domain) and stress as a function of parent characteristics (e.g., depression, sense of competence, social isolation; Parent Domain), as well as an overall stress score (Total Stress). Raw scores are calculated (normative means: Child Doman = 98.4; Parent Domain = 122.7; Total Stress Score = 221.1). This measure was given at all time points. Scores range from 131-320 for Total Stress, 69-188 for Parent Domain, and 50-145 for Child Domain, with higher scores indicative of greater stress (Total: >260; Parent: >153, Child: >122).
Time Frame: Baseline (at study entry), 6 months, 1 year, 2 years, 3 years, and 5 years
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | 6 Months | 1 Year | 2 Years | 3 Years | 5 Years
Number analyzed (Participants) | 25 | 30 | 50 | 64 | 67 | 60
units on a scale
  Child Domain | 96.76 (20.91) | 93.08 (15.98) | 93.27 (14.86) | 92.77 (16.23) | 94.60 (18.69) | 92.49 (19.02)
  Parent Domain | 109.38 (30.33) | 101.56 (22.90) | 105.84 (22.90) | 105.84 (27.56) | 105.92 (24.96) | 102.74 (24.97)
  Overall Total Stress | 207.25 (47.07) | 194.84 (23.36) | 200.51 (35.98) | 198.61 (38.52) | 200.23 (40.21) | 194.68 (39.84)

25. Secondary Outcome: Assessment of School Readiness
Description: The Bracken Basic Concepts Scale was used to assess school readiness. It is an examiner-administered measure that assesses per-academic skills including letter and number recognition, shapes, colors, and understanding of sizes and comparisons. Raw scores are converted into age-normed scaled scores (normative mean = 10, SD = 3) for the School Readiness Composite. Higher scores are indicative of stronger pre-academic skills, with scores from 7 to 13 within the Average range.
Time Frame: Patients were assessed at 5 years of age
Population: All patients were included, regardless of treatment strata.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 5 Years
Number analyzed (Participants) | 60
units on a scale | 8.96 (3.10)

26. Secondary Outcome: Number of Participants With Development of Pineal Cysts
Description: The MRI reports from bilateral patients were reviewed and data abstracted regarding pineal gland measurement and information about pineal cysts. The number of participants with change in primary visual cortex function from diagnosis through 6 years after last patient enrollment is reported here.
Time Frame: At diagnosis through 6 years after last patient enrollment
Population: A patient may be included in more than one category due to having more than one cyst.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Bilateral Retinoblastoma: Results were analyzed for all participants regardless of stratum. All participants received chemotherapy (5 Stratum C, high risk; 11 Stratum A; 27 Stratum B).
Arm/Group | Participants With Bilateral Retinoblastoma
Number analyzed (Participants) | 43
Participants
  Developed new solitary cyst(s) | 12
  Developed multiple new cysts | 15
  Growth of pineal cyst | 5
  Decrease in size (resolution) of pineal cyst | 1
  No change | 11

27. Secondary Outcome: Number of Participants With Change in Size of Pineal Gland
Description: The MRI reports from bilateral patients were reviewed and data abstracted regarding pineal gland measurement and information about pineal cysts. The number of participants with change in pineal gland size is reported here.
Time Frame: From diagnosis through 6 years after last patient enrollment
Population: Pineal gland size was measured during routine MRI screening. Measurements were compared over time to quantify any change in size. Measurements were compared with standard pediatric norms to determine "prominence" or "mild enlargement" (subjective comparison).
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Bilateral Retinoblastoma
Number analyzed (Participants) | 43
Participants
  Prominent or mildly enlarged pineal glands | 12
  Pineal growth over time | 8
  No change in pineal gland size | 23

28. Secondary Outcome: Change in Distortion Product Otoacoustic Emissions (DPOAEs)
Description: For DP_amplitude to be considered valid, a baseline DP_SNR (Distortion Product for Signal-to-noise ratio) for each frequency (1000-8000 Hz) and for each ear (left and right) must be = 6 dB. Any ear with invalid amplitude at baseline for each frequency should be excluded. The DPOAEs amplitude levels were averaged across the right and left ears at each frequency in the patients exhibiting valid DPOAE amplitudes in both ears, resulting in mean DPOAE levels. Subsequently, comparisons between baseline and most recent evaluation (collapsed across ears) for each frequency were made to evaluate if a significant decrease in DPOAE amplitude exists between the two time points.
Time Frame: From Diagnosis through 5 years after completion of therapy
Population: A total of 14 patients had "Incomplete data" and were not included in the analysis.
Measure: Mean (Standard Deviation); unit: dB
Groups:
- Baseline; Interim Evaluation; Additional Evaluation: All Stratum B participants with non-missing observation values were included. Stratum B (Advanced Bilateral retinoblastoma) includes patients with at least one Reese-Ellsworth group IV or V eye that after careful evaluation by the treating team is considered not to require upfront enucleation. A proportion of patients treated on this stratum will not have advanced disease in both eyes. Only stratum B patients received window therapy consisting of 2 courses of vincristine and topotecan.
Arm/Group | Baseline | Interim Evaluation | Additional Evaluation
Number analyzed (Participants) | 13 | 12 | 4
dB
  1000 Hz: number analyzed (Participants) | 3 | 12 | 4
  1000 Hz | 17.7 (16.6) | 5.5 (2.5) | 4.5 (1.7)
  1400 Hz: number analyzed (Participants) | 6 | 12 | 4
  1400 Hz | 16.6 (3.6) | 9.4 (2.5) | 8.2 (2.8)
  2000 Hz: number analyzed (Participants) | 11 | 12 | 4
  2000 Hz | 15.1 (1.7) | 13.0 (1.8) | 11.0 (1.4)
  2800 Hz | 11.6 (2.0) | 12.2 (1.9) | 8.4 (3.2)
  4000 Hz | 15.3 (4.8) | 11.3 (1.9) | 3.4 (6.6)
  6000 Hz | 13.3 (2.0) | 12.9 (2.2) | 5.7 (8.6)
  8000 Hz: number analyzed (Participants) | 12 | 12 | 4
  8000 Hz | 5.0 (1.9) | -2.0 (3.2) | -9.9 (6.0)

29. Secondary Outcome: Mean Primary Visual Cortex Function: Cluster Size
Description: Functional magnetic resonance imagining (fMRI) was used to investigate primary visual cortex (V1) response to visual stimulation in 105 children being treated for intraocular retinoblastoma. Primary visual cortex activity was assessed in each subject using blood oxygenation level-dependent (BOLD) signal. The BOLD signal was analyzed via a general linear model using Statistical Parametric Mapping software (SPM, Wellcome Institute of Neuology, London).
  Voxel volume/peak BOLD response is a measurement of the volume of activation of the cortex. There is no known association with visual outcome at this time.
Time Frame: At diagnosis through 6 years after last patient enrollment
Measure: Mean (Standard Deviation); unit: number activated voxels (negative BOLD)
Units Other Than Participants: Number of exams
Arm/Group | Stratum A | Stratum B | Stratum C
Number analyzed (Participants) | 12 | 24 | 41
Number analyzed (Number of exams) | 33 | 152 | 122
number activated voxels (negative BOLD) | 2372 (2640) | 1080 (2916) | 2105 (2476)

30. Post Hoc Outcome: Number of Patients Recommended for and Utilizing Rehabilitation Services
Description: Participants were evaluated by Occupational Therapy at diagnosis, and at 3, 6, 9, and 12 months from diagnosis with a battery of standardized and non-standardized measures. Assessments including the Battelle Developmental Inventory, the Sensory Profile, the Oregon Project for Visually Impaired Preschoolers, Pediatric Evaluation of Disability Inventory, and the Greenspan Social Emotional Growth Scale were utilized for developing the participants plan of care and making referrals for services in the home community. Recommendations for rehabilitation services in the home community were made based on the results of the occupational therapists evaluation.
  A subsequent review of February 2013 subgroup definitions resulted in the reclassification of evaluable participants and subgroups in May 2015. This reclassification applies to the data for this outcome only.
Time Frame: At diagnosis, and at 3, 6, 9, and 12 months from diagnosis
Population: Objective was added after the protocol started. Due to the late start, 33 of the 105 overall participants were eligible. Of the 33, 1 family declined to participate; 1 was removed from the protocol, 5 were lost to follow-up, and 4 patients were unable to complete the developmental assessment. In total, 22 have complete data sets.
Measure: Number; unit: participants
Groups:
- Occupational Therapy Recommended Rehabilitation Services: Occupational therapy evaluation recommended rehabilitation services.
- Occupational Therapy Did Not Recommend Rehabilitation Services: Occupational therapy evaluation did not recommend rehabilitation services.
Arm/Group | Occupational Therapy Recommended Rehabilitation Services | Occupational Therapy Did Not Recommend Rehabilitation Services
Number analyzed (Participants) | 16 | 6
participants
  Received rehabilitation services | 12 | 1
  Did not receive rehabilitation services | 4 | 5

31. Secondary Outcome: Mean Primary Visual Cortex Function: Maximum T-value
Description: Functional magnetic resonance imagining (fMRI) was used to investigate primary visual cortex (V1) response to visual stimulation in 105 children being treated for intraocular retinoblastoma. Primary visual cortex activity was assessed in each subject using blood oxygenation level-dependent (BOLD) signal. The BOLD signal was analyzed via a general linear model using Statistical Parametric Mapping software (SPM, Wellcome Institute of Neurology, London). The maximum t-statistic in activated cluster (negative BOLD) is provided.
  Voxel volume/peak BOLD response is a measurement of the volume of activation of the cortex. There is no known association with visual outcome at this time.
Time Frame: At diagnosis through 6 years after last patient enrollment
Measure: Mean (Standard Deviation); unit: Maximum t-statistic (negative BOLD)
Units Other Than Participants: Number of exams
Arm/Group | Stratum A | Stratum B | Stratum C
Number analyzed (Participants) | 12 | 24 | 41
Number analyzed (Number of exams) | 33 | 152 | 122
Maximum t-statistic (negative BOLD) | 7.9 (6.9) | 6.2 (3.9) | 8.8 (4.7)

ADVERSE EVENTS:
Time Frame: Adverse events have been collected from study activation (February 2005) through June, 2011.
Arm/Group | Stratum A | Stratum B | Stratum C
Serious Adverse Events (participants affected / at risk) | 1/23 | 9/27 | 1/55
Other Adverse Events (participants affected / at risk) | 23/23 | 27/27 | 18/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A (N=23) | Stratum B (N=27) | Stratum C (N=55)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 8 (9) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hearing: patients with/without baseline audiogram and enrolled in a monitoring program (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils, colon (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils, cellulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum A (N=23) | Stratum B (N=27) | Stratum C (N=55)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 23 (161) | 26 (271) | 18 (69)
Platelets (Blood and lymphatic system disorders) | 9 (22) | 25 (86) | 10 (32)
Hemoglobin (Blood and lymphatic system disorders) | 10 (22) | 23 (72) | 14 (34)
Leukocytes (Blood and lymphatic system disorders) | 3 (5) | 20 (36) | 14 (23)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented) (Infections and infestations) | 2 (3) | 17 (30) | 3 (3)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils, upper airway (Infections and infestations) | 2 (2) | 4 (4) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils, cellulitis (Infections and infestations) | 1 (2) | 4 (4) | 0 (0)
Infection(documented clinically or microbiologically with Grade 3 or 4 neutrophils,catheter-related (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils, Catheter-related (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (Infections and infestations) | 0 (0) | 8 (8) | 0 (0)
Anorexia (Gastrointestinal disorders) | 1 (1) | 6 (9) | 0 (0)
Dehydration (Gastrointestinal disorders) | 3 (4) | 5 (5) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 7 (10) | 1 (1)
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5) | 2 (2) | 1 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (8) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes